CLINICAL TRIAL: NCT05249439
Title: Investigation of a New Diet for the Treatment of Obesity in the NHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16HH3487; 189449 (Other: Integrated Research Approval System (IRAS)); 16/LO/1622 (Other: Research Ethics Committee (REC) reference)
Record Dates: First submitted 2021-11-22; First posted 2022-02-21 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: Obesity, Tier 3, weight-loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Two groups of patients will be recruited from our hospital obesity clinic. One group will take part in the I-SatPro weight management programme One group will take part in the Tier 3 weight loss programme that is currently offered in our clinical service.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-SatPro (Experimental): Patients in the I-SatPro group will attend I-SatPro patient group weight management sessions (Tier 3 equivalent) and follow the I-SatPro programme
  Interventions: Other: I-SatPro weight loss programme
- Control (Active Comparator): Patients in the control group will attend the established Imperial Weight Centre Tier 3 patient group weight management sessions and follow the Imperial Weight Centre Tier 3 weight management programme
  Interventions: Other: Tier 3 weight loss programme

INTERVENTIONS:
Other: I-SatPro weight loss programme — I-SatPro weight loss programme: participants advised on I-SatPro dietary change as well as eating patterns, lifestyle change such as exercise, self-care such as advice on sleep and behavioural change strategies.
  Arms: I-SatPro
Other: Tier 3 weight loss programme — Tier 3 weight loss programme: participants advised to make changes to food choices in accordance with NHS healthy eating advice, eating habits, lifestyle change such as exercise, mindful eating and behavioural change strategies.
  Arms: Control

SUMMARY:
Over one in four adults living in the UK is living with obesity. Obesity is associated with health complications including type 2 diabetes, heart disease and depression. The current NHS treatment for obesity includes attending a specialist hospital weight management service called 'Tier 3' where patients receive help from healthcare professionals such as doctors, dieticians and psychologists. It is known that health conditions associated with obesity improve or reverse if a person with obesity loses five per cent or more of their body weight. On average, currently available Tier 3 programmes achieve less weight loss than this. In our specialist obesity clinic at the Imperial Weight Centre, we (the study research team) have designed a new weight loss programme called Imperial Satiety Protocol (or I-SatPro for short). I-SatPro comprises dietary advice including eating a low carbohydrate (low glycaemic index) diet, eating protein for the satiating effects, eating healthy fats and abstaining from high sugar and/or processed foods which can drive over-eating. Participants will be advised to eat according to subjective feelings of hunger and fullness, rather than eating according to a defined calorie restriction. Similar to other Tier 3 Programmes, I-SatPro also contains locally devised content related to healthy eating, for example fibre intake, the timing of eating, lifestyle change such as exercise, self-care such as advice on sleep and behavioural change strategies.

DETAILED DESCRIPTION:
The purpose of this feasibility/pilot study is to check whether:

1. Our patients like I-SatPro
2. Whether our patients want to follow I-SatPro
3. Check whether our patients following I-SatPro achieve improvements in their health including: weight loss, changes in blood pressure, changes in diabetes control, changes in blood lipids 'cholesterol', changes in their eating patterns and relationship with food, changes in their wellbeing

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Male or female
* Body mass index ≥35kg/m2 with at least one obesity related co-morbidity
* Body mass index ≥40kg/m2 with or without an obesity related co-morbidity
* Eligible for treatment under the NHS

Exclusion Criteria:

* History of any medical, psychological or other condition, or use of any medications, which would either compromise the validity of the study or the safety of the participant
* English language fluency and comprehension insufficient to be able to participate in educational and group components of the programme
* Usual residence/place of work is sufficiently far from the study site or logistical/lifestyle factors mean that it is likely that the patient would be unable to attend for all sessions/components of the study
* Pregnancy or breast feeding
* Previous bariatric surgery
* Concurrent participation in another research study which would either compromise the validity of the study or the safety of the participant
* Previous participation in a study if the investigators judge that this would either compromise the validity of the study or the safety of the participant
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tricia Tan, MBChB, PhD, Principal Investigator — Imperial College London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hameed S, Salem V, Alessimii H, Scholtz S, Dar O, Miras AD, Meeran K, Bloom SR, Ahmed AR, Purkayastha S, Chahal H, Tan T. Imperial Satiety Protocol: A new non-surgical weight-loss programme, delivered in a health care setting, produces improved clinical outcomes for people with obesity. Diabetes Obes Metab. 2021 Jan;23(1):270-275. doi: 10.1111/dom.14207. Epub 2020 Oct 15. PMID 32991078

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants in the I-SatPro group were excluded for the following reasons: psychiatric (n=1), medical (n=1), literacy (n=1) Two participants dropped out. Ten participants in the I-SatPro arm completed the study. Primary outcome data were available for: n=10 Zero participants in the control arm completed the study.
Groups:
- I-SatPro: Patients in the I-SatPro group will attend I-SatPro patient group sessions and follow the I-SatPro weight loss programme
- Control: Patients in the control group will attend established NHS Tier 3 patient group sessions (standard care) and follow the NHS Tier 3 weight loss programme
Period: Overall Study
Arm/Group | I-SatPro | Control
Started | 15 | 6
Completed | 10 (Three participants in the I-SatPro group were excluded for the following reasons: psychiatric (n=1), medical (n=1), literacy (n=1) Two participants dropped out. Ten participants in the I-SatPro arm completed the study.) | 0 (Five participants dropped out. As the intervention was dietary advice to patients delivered in a group setting it was not feasible to continue this arm of the intervention with one patient remaining. This remaining participant (one patient) was therefore withdrawn by physician decision. Zero participant completed this arm of the study.)
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Physician Decision | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | I-SatPro | Control | Total
Number analyzed (Participants) | 15 | 6 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 6 | 20
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.5 (8.6) | 42.8 (14.4) | 43.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 6 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 1 | 6
  South Asian | 5 | 2 | 7
  Middle Eastern | 2 | 1 | 3
  Black (Caribbean) | 1 | 1 | 2
  Black (African) | 1 | 0 | 1
  Asian (other) | 0 | 1 | 1
  Mixed | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 15 | 6 | 21
Weight units: kg [Mean (Standard Deviation); unit: kg] | 112.8 (24.0) | 133.1 (24.1) | 118.6 (25.2)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 41.3 (9.4) | 45.3 (6.0) | 42.4 (8.6)

OUTCOME MEASURES:

1. Primary Outcome: Body Weight Change
Description: Change in body weight will be measured from patient group session 1 (week 0) to the end of study (week 52)
Time Frame: First patient group visit (week 0) to end of study (week 52)
Population: Baseline pre-dietary intervention and post-dietary intervention (week 52) data were available for n=10 participants in the I-SatPro group and body weight change was analyzed in these participants.
  No patients were analysed for the control group: it was not possible to analyze change in body weight for the control group at the end of the study (week 52) as these data were not collected because no participants remained in this arm of the study at this timepoint.
Measure: Mean (Standard Error); unit: kg
Groups:
- Control: Patients in the control group will attend established NHS Tier 3 patient group sessions (standard clinical care) and follow the Imperial Weight Centre Tier 3 weight loss programme
Arm/Group | I-SatPro | Control
Number analyzed (Participants) | 10 | 0
kg | -12.99 (1.7) |
Statistical Analysis 1: Comparison: I-SatPro; I-SatPro starting weight Vs 52 week weight (kg); Test type: Other — Paired t-test; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -12.99

2. Secondary Outcome: Energy Expenditure (How Efficiently Your Body Burns Calories)
Description: Measurement of whether the dietary intervention changes the rate at which your body burns calories
Time Frame: Pre-dietary intervention (baseline) and end of study post-dietary intervention (week 52)
Population: Resting energy expenditure corrected for body weight (kcal/kg)
  In analysis of this secondary outcome measure:
  Baseline pre-dietary intervention and post-dietary intervention (week 52) data were available for n=9 participants in the I-SatPro group.
  Baseline data were available for n=4 out of 6 participants in the control group. No data were collected for the week 52 time point: data were available for n=0 participants post-dietary intervention (week 52) (please see pre-assignment details).
Measure: Mean (Standard Error); unit: kcal/kg
Arm/Group | I-SatPro | Control
Number analyzed (Participants) | 9 | 4
kcal/kg
  Resting energy expenditure corrected for body weight (kcal/kg) pre-intervention (baseline) | 17.8 (1.4) | 17.7 (0.8)
  Resting energy expenditure corrected for body weight (kcal/kg) post-dietary intervention (week 52): number analyzed (Participants) | 9 | 0
  Resting energy expenditure corrected for body weight (kcal/kg) post-dietary intervention (week 52) | 18.0 (0.6) |

3. Secondary Outcome: Body Weight Composition - How Much of Your Weight is Body Fat?
Description: Percentage body fat as measured using bio-impedance weighing scales
  Although baseline data were recorded by the study team, inter-individual differences at the same timepoint indicated recorded measure of insufficient reliability to continue to record/report.
Time Frame: Pre-dietary intervention (baseline) and post-dietary intervention (week 52)
Population: Participant baseline data are reported. One participant in the Control group was unable to comply with instructions for bio-impedance scale use
Measure: Mean (Standard Error); unit: Percentage body fat (%)
Arm/Group | I-SatPro | Control
Number analyzed (Participants) | 9 | 5
Percentage body fat (%) | 43.8 (2.3) | 48.7 (2.9)

4. Secondary Outcome: Change in Blood Pressure
Description: Measuring patients' blood pressure to see if it changes
Time Frame: Pre-dietary intervention (baseline) and end of study post-dietary intervention (week 52)
Population: Baseline pre-dietary intervention and post-dietary intervention (week 52) data were available for n= 9 participants in the I-SatPro group and change in blood pressure was analyzed in these participants.
  No patients were analysed for the control group: it was not possible to analyze change in blood pressure for the control group at the end of the study (week 52) as these data were not collected because no participants remained in this arm of the study at this timepoint.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | I-SatPro | Control
Number analyzed (Participants) | 9 | 0
mmHg | -6.0 (3.7) |

5. Secondary Outcome: Change in Blood Sugar Levels (Changes in the Blood Test Marker for Diabetes Called HbA1c)
Description: Change in blood sugar levels measured using the blood test marker for diabetes (glycemic control) called HbA1c
Time Frame: Pre-dietary intervention (baseline) and end of study post-dietary intervention (week 52)
Population: Baseline pre-dietary intervention and post-dietary intervention (week 52) data were available for n=9 participants in the I-SatPro group and change in HbA1c was analyzed in these participants.
  No patients were analysed for the control group: it was not possible to analyze change in HbA1c for the control group at the end of the study (week 52) as these data were not collected because no participants remained in this arm of the study at this timepoint.
Measure: Mean (Standard Error); unit: mmol/mol
Arm/Group | I-SatPro | Control
Number analyzed (Participants) | 9 | 0
mmol/mol | -1.3 (1.0) |

6. Secondary Outcome: Measurement of Eating Patterns, Hunger Levels and Relationship With Food
Description: Three Factor Hunger Questionnaire:
  The TFEQ is a 51-item questionnaire completed by study participants to measure three areas (or factors) related to eating behaviour: cognitive restraint of eating (score 0 to 20), disinhibition (score 0 to 16), and hunger (score 0 to 15).
  The higher the score the greater the level of restrained eating, disinhibited eating and subjective feelings of/predisposition to feeling hungry.
Time Frame: Pre-dietary intervention (baseline) and post-dietary intervention (week 52)
Population: In analysis of this secondary outcome measure:
  In the I-SatPro group: a set of baseline and week 52 data were available for n=7 participants No data were collected for the week 52 time point: in the control group baseline data were available for n=6 participants and post-dietary intervention (week 52) data were available for n=0 participants (please see pre-assignment details).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | I-SatPro | Control
Number analyzed (Participants) | 7 | 6
Score on a scale
  Hunger score pre-dietary intervention | 8.4 (4.6) | 6.8 (3.1)
  Hunger score post-intervention: number analyzed (Participants) | 7 | 0
  Hunger score post-intervention | 0.7 (0.5) |
  Cognitive restraint of eating pre-dietary intervention | 10.0 (2.6) | 9.7 (4.8)
  Cognitive restraint of eating post-dietary intervention: number analyzed (Participants) | 7 | 0
  Cognitive restraint of eating post-dietary intervention | 10.4 (4.0) |
  Disinhibition score pre-dietary intervention | 11.1 (3.4) | 8.5 (4.2)
  Disinhibition score post-dietary intervention: number analyzed (Participants) | 7 | 0
  Disinhibition score post-dietary intervention | 4.0 (2.0) |

7. Secondary Outcome: Change in Scores Across the Three Measured Domains (Emotional Eating, External Eating and Restrained Eating) on Dutch Eating Behaviours Questionnaire (DEBQ)
Description: The DEBQ questionnaire completed by study participants to assess eating behaviour across three domains:
  Emotional eating - eating in response to negative emotions External eating - eating in response to external cues such as the sight or smell of food Restrained eating - the conscious limiting of food intake The DEBQ consists of 33 items grouped into the three categories: emotional eating (13 items), external eating (10 items) and restrained eating (10 items) Participant responses to each item range from 1 (never) to 5 (very often) with higher scores indicating a greater endorsement of the eating behaviour described in the question.
  The lowest total score for the DEBQ (combined for all three categories) is 33 indicating no behaviours relating to the three domains eating and the highest score is 165 indicating very frequent behaviours relating to the three domains. A lower score indicates healthy eating behaviours, a higher score indicates more problematic eating behaviours.
Time Frame: Pre-dietary intervention (baseline) and post-dietary intervention (week 52)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | I-SatPro | Control
Number analyzed (Participants) | 7 | 6
Score on a scale
  Total score restrained eating (baseline) Scale range: Minimum score: 10 Maximum score: 50 | 27.3 (4.2) | 32.8 (7.2)
  Total score restrained eating (week 52) Scale range: Minimum score: 10 Maximum score: 50: number analyzed (Participants) | 7 | 0
  Total score restrained eating (week 52) Scale range: Minimum score: 10 Maximum score: 50 | 33.4 (8.8) |
  Total score emotional eating (baseline) Scale range: Minimum score: 13 Maximum score: 65 | 53.3 (11.2) | 35.8 (17.6)
  Total score emotional eating (week 52) Scale range: Minimum score: 13 Maximum score: 65: number analyzed (Participants) | 7 | 0
  Total score emotional eating (week 52) Scale range: Minimum score: 13 Maximum score: 65 | 28.3 (10.5) |
  Total score external eating (baseline) Scale range: Minimum score: 10 Maximum score: 50 | 34.1 (7.0) | 30.5 (6.4)
  Total score external eating (week 52) Scale range: Minimum score: 10 Maximum score: 50: number analyzed (Participants) | 7 | 0
  Total score external eating (week 52) Scale range: Minimum score: 10 Maximum score: 50 | 19.3 (5.8) |

8. Secondary Outcome: Measurement of Wellbeing and Quality of Life
Description: This secondary outcome measures will be assessed using the Short Form-36 (SF-36) questionnaire.
  SF-36 is a participant completed questionnaire consisting of 36 questions relating to quality of life and well-being.
  Questions cover the following eight domains:
  Physical functioning Role limitation due to physical health Role limitation due to emotional problems Energy/fatigue Emotional wellbeing Social functioning Pain General Health
  Each of these domains is scored from 0 to 100 with a higher score indicating better quality of life and well-being.
Time Frame: Pre-dietary intervention (baseline) and post-dietary intervention (week 52)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | I-SatPro | Control
Number analyzed (Participants) | 7 | 6
Score on a scale
  SF-36 score physical functioning pre-dietary intervention (baseline) out of 100 | 70.0 (16.8) | 45 (30.7)
  SF-36 score physical functioning post-dietary intervention (week 52) out of 100: number analyzed (Participants) | 7 | 0
  SF-36 score physical functioning post-dietary intervention (week 52) out of 100 | 98.6 (2.4) |
  SF-36 score role limitation due to physical health pre-dietary intervention (baseline) out of 100 | 53.6 (46.6) | 25.0 (38.7)
  SF-36 score role limitation due to physical health post-dietary intervention (week 52) out of 100: number analyzed (Participants) | 7 | 0
  SF-36 score role limitation due to physical health post-dietary intervention (week 52) out of 100 | 100 (0) |
  SF-36 score role limitation due to emotional problems pre-dietary intervention (baseline) out of 100 | 76.2 (31.7) | 27.8 (39.0)
  SF-36 score role limitation due to emotional problems post-dietary intervention (week 52) out of 100: number analyzed (Participants) | 7 | 0
  SF-36 score role limitation due to emotional problems post-dietary intervention (week 52) out of 100 | 95.2 (12.6) |
  SF-36 score energy/fatigue pre-dietary intervention (baseline) out of 100 | 47.1 (13.8) | 37.5 (16.4)
  SF-36 score energy/fatigue post-dietary intervention (week 52) out of 100: number analyzed (Participants) | 7 | 0
  SF-36 score energy/fatigue post-dietary intervention (week 52) out of 100 | 86.4 (9.0) |
  SF-36 score emotional wellbeing pre-dietary intervention (baseline) out of 100 | 67.4 (15.4) | 56.7 (9.9)
  SF-36 score emotional wellbeing post-dietary intervention (week 52) out of 100: number analyzed (Participants) | 7 | 0
  SF-36 score emotional wellbeing post-dietary intervention (week 52) out of 100 | 89.7 (6.0) |
  SF-36 score social functioning pre-dietary intervention (baseline) out of 100 | 62.5 (26.0) | 58.3 (25.8)
  SF-36 score social functioning post-dietary intervention (week 52) out of 100: number analyzed (Participants) | 7 | 0
  SF-36 score social functioning post-dietary intervention (week 52) out of 100 | 98.2 (4.7) |
  SF-36 score pain pre-dietary intervention (baseline) out of 100 | 67.5 (29.9) | 44.6 (18.5)
  SF-36 score pain post-dietary intervention (week 52) out of 100: number analyzed (Participants) | 7 | 0
  SF-36 score pain post-dietary intervention (week 52) out of 100 | 92.5 (12.0) |
  SF-36 score general health pre-dietary intervention (baseline) out of 100 | 47.1 (26.1) | 31.7 (18.1)
  SF-36 score general health post-dietary intervention (week 52) out of 100: number analyzed (Participants) | 7 | 0
  SF-36 score general health post-dietary intervention (week 52) out of 100 | 85.0 (8.2) |

9. Secondary Outcome: Patient Drop-out Rate
Description: Patient drop out will be recorded. Drop out will be defined as a patient expressing the wish to drop out either verbally or in writing. A patient will also be considered to have dropped out of the study if they do not attend patient group sessions or fail to attend study visits without providing the investigators with an explanation for their non-attendance. Drop-out rate will be used as a surrogate marker of the acceptability of the intervention to patients.
Time Frame: Patient drop out will be recorded from the first patient group session (week 0) to the end of the study (week 52).
Measure: Count of Participants; unit: Participants
Arm/Group | I-SatPro | Control
Number analyzed (Participants) | 15 | 6
Participants | 2 | 5

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | I-SatPro | Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/6
Other Adverse Events (participants affected / at risk) | 0/15 | 0/6

LIMITATIONS AND CAVEATS:
The dropout rate in the control group (standard Tier 3 care) was too high to feasibly continue this arm of the study.

Technical problems with measurement of percentage body fat resulted in unreliable and uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT05249439/Prot_SAP_000.pdf